CLINICAL TRIAL: NCT06551441
Title: Cardiopulmonary Adaptations to High-intensity Interval Training (HIIT) in COPD: a Randomized Controlled Trial (the COPDEX Study)
Brief Title: Cardiopulmonary Adaptations to High-intensity Interval Training (HIIT) in COPD
Acronym: COPDEX
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Ronan Berg, MD, DMSc, Associate Professor, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-24021751
Record Dates: First submitted 2024-06-19; First posted 2024-08-13 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: COPD; Rehabilitation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — High-Intensity Interval Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise (Experimental): The HIIT intervention includes three supervised sessions per week over a 24-week period i.e., 72 exercise sessions and take place at CFAS or at home with supervision
  Interventions: Behavioral: High Intensity Interval Training (HIIT)
- Control group (No Intervention): Controls will be encouraged to maintain current exercise habits for the duration of the study.

INTERVENTIONS:
Behavioral: High Intensity Interval Training (HIIT) — The HIIT intervention consist of 4 intervals with each lasting 4 minutes (4x4min). If a participant reports discomfort related to the length of the intervals or start to feel unmotivated by performing the same exercise, we will use another HIIT protocol: 10x1min.
  The 4x4min HIIT consists of a warm-up period of 10 minutes with a target heart rate at 60-70% of HRmax, followed by 4 HIIT intervals with a target HR ≥85%. The intervals are separated by three minutes of active rest, in which the HR should drop to 60% of maximum. Following this, a cool down period of three minutes at warm up intensity is performed.
  The 10x1min HIIT consists of a 10-minute warm-up period.The warm-up is followed by 10 intervals, each lasting 1 min at 100% of maximal workload, separated by three minutes of active rest, in which the HR should drop to 60% of maximum. Following the intervals, a cool down period of three minutes at warm up intensity is performed.
  Arms: Exercise

SUMMARY:
The aim of this prospective randomised controlled trial in which the impact of high intensity interval training (HIIT) on pulmonay blood volume, pulmonary gas exchange during exercise, and lung tissue mass.

The primary objective is to investigate whether 6 months of supervised HIIT leads to an increase in pulmonary blood volume in patients with COPD with a concomitant improvement in pulmonary gas exchange.

Key objectives are to determine whether an increase in pulmonary blood volume is associated with the formation of new lung tissue. Other secondary objectives include investigating the effect of supervised HIIT on formation of lung tissue, symptom severity, pulmonary gas exchange at supine rest and on pulmonary blood volume at rest. Finally, exploratory objectives include investigating the effects of HIIT on lung function, V̇O2peak, functional outcomes, body composition, blood samples and cardiac output.

Participants will be randomly allocated (1:1) stratified by sex to either

1. 24 weeks of HIIT training consisting of 3 weekly supervised exercise sessions or
2. A control group who will not undergo HIIT training. The control group will be encouraged not to change their exercise or eating habits.

The participants will visit the clinic pre- and post the intervention. Exercise habits, adverse events, hospital admisseions, infections and medications will be assessed by phone at week 4, 8, 12, 16, 20 and at follow-up visit. All participants will undergo 24-h accelerometry for five consecutive days to measure posture allocation and daily physical activity behavior. The devices will be attached just before the randomization, after one month, at 12 weeks and just before the 6 months testing.

ELIGIBILITY:
Inclusion criteria

* Men and women
* Age >=40 and <80 years
* COPD (GOLD stage I to III)
* Modified Medical Research Council score (mMRC) of 0 to 3
* Resting arterial oxygenation > 90% Exclusion criteria
* Symptoms of ischaemic heart disease
* Known heart failure
* Unable to complete or understand HIIT training
* Claudication
* Symptoms of disease within 2 weeks prior to the study
* Participation in pulmonary rehabilitation within 3 months
* Known malignant disease
* Pregnancy
* Unstable cardiac arrhythmic disease
* Renal or liver dysfunction

  * Known chronic kidney or liver disease
  * Elevated creatinine, urea, alanine transaminase (ALAT), aspartate transaminase (ASAT), bilirubin, basic phosphatases at blood test
* Completion of pulmonary rehabilitation within the last 3 months

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Pulmonary blood volume (mL) at rest | 6 months
  Difference in change from baseline to six months between groups in pulmonary blood volume (mL) at rest

SECONDARY OUTCOMES:
DL,NO (mmol/(min kPa)) as a function of V̇O2 measured at rest | 6 months
  Difference in change from baseline to six months between groups in DL,NO (mmol/(min kPa)) as a function of V̇O2 measured at rest, 60% of current maximal workload (relative), and at follow-up including 60% of maximal workload at baseline (absolute)
Total LTM (g) | 6 months
  Difference in change from baseline to six months between groups in total LTM (g)

OTHER OUTCOMES:
DL,NO (mmol/(min kPa)) during exercise at 60% of current maximal workload (relative) | 6 months
  Difference in change from baseline to six months between groups in DL,NO (mmol/(min kPa)) during exercise at 60% of current maximal workload (relative)
DL,NO (mmol/(min kPa)) during exercise at 60% of the maximal workload measured at baseline (absolute) | 6 months
  Difference in change from baseline to six months between groups in DL,NO (mmol/(min kPa)) during exercise at 60% of the maximal workload measured at baseline (absolute)
Pulmonary blood volume / total blood volume ratio | 6 months
  Difference in change from baseline to six months between groups in pulmonary blood volume / total blood volume ratio
Health-related quality of life - COPD Assessment Test (CAT) score | 6 months
  Difference in change from baseline to six months between groups in health-related quality of life
Health-related quality of life - St. George's Respiratory Questionnaire (SGRQ) | 6 months
  Difference in change from baseline to six months between groups in health-related quality of life
Lobar LTM (g) | 6 months
  Difference in change from baseline to six months between groups in lobar LTM (g)
LTM/1.73 m2 BSA (g/m2) | 6 months
  Difference in change from baseline to six months between groups in LTM/1.73 m2 BSA (g/m2)
Total blood volume | 6 months
  Difference in change from baseline to six months between groups in total blood volume
DL,NO (mmol/(min kPa)) during upright rest | 6 months
  Difference in change from baseline to six months between groups in DL,NO (mmol/(min kPa)) during upright rest
DL,CO,5s (mmol/(min kPa)) during upright rest | 6 months
  Difference in change from baseline to six months between groups in DL,CO,5s (mmol/(min kPa)) during upright rest
Pulmonary capillary blood volume (VC, mL) during upright rest | 6 months
  Difference in change from baseline to six months between groups in pulmonary capillary blood volume (VC, mL) during upright rest
Alveolar-capillary membrane diffusing capacity (DM, mmol/(min kPa)) during upright rest | 6 months
  Difference in change from baseline to six months between groups in alveolar-capillary membrane diffusing capacity (DM, mmol/(min kPa)) during upright rest
DL,NO (mmol/(min kPa)) during supine rest | 6 months
  Difference in change from baseline to six months between groups in DL,NO (mmol/(min kPa)) during supine rest
DL,CO,5s (mmol/(min kPa)) during supine rest | 6 months
  Difference in change from baseline to six months between groups in DL,CO,5s (mmol/(min kPa)) during supine rest
Pulmonary capillary blood volume (VC, mL) during supine rest | 6 months
  Difference in change from baseline to six months between groups in pulmonary capillary blood volume (VC, mL) during supine rest
Alveolar-capillary membrane diffusing capacity (DM, mmol/(min kPa)) during supine rest | 6 months
  Difference in change from baseline to six months between groups in alveolar-capillary membrane diffusing capacity (DM, mmol/(min kPa)) during supine rest
Cardiac output (L/min) during exercise | 6 months
  Difference in change from baseline to six months between groups in cardiac output (L/min) during exercise at 60% of current maximal workload and 60% of baseline maximal workload, in the supine position, and during upright rest
DL,CO,NO-based V̇O2 during exercise | 6 months
  DL,CO,NO-based V̇O2 during exercise at 60% of current maximal workload and 60% of baseline maximal workload, in the supine position, and during upright rest
V̇O2peak | 6 months
  Difference in change from baseline to six months between groups in relative (mL/kg/min) and absolute (mL/min) V̇O2peak, ventilatory threshold (%), and ventilatory reserve (%)
Time constant (s) | 6 months
  Difference in change from baseline to six months between groups in time constant from V̇O2kinetic test
Amplitude (ml/kg^-1/min^-1) | 6 months
  Difference in change from baseline to six months between groups in amplitude measured by V̇O2kinetic test
Time delay (s) | 6 months
  Difference in change from baseline to six months between groups in time delay measured by V̇O2kinetic test
Hand-grip strength (kg) | 6 months
  Difference in change from baseline to six months between groups in hand-grip strength (kg)
Sit-to-stand test (n) | 6 months
  Difference in change from baseline to six months between groups in numbers of completed 30 seconds sit-to-stand test (n)
Body composition: | 6 months
  Difference in change from baseline to six months between groups in body composition: total mass (kg), total fat mass (kg and %), lean body mass (kg), fat percentage (%)
Lung function | 6 months
  Difference in change from baseline to six months between groups in lung function: FEV1 (L and %pred), FVC (L and %pred), RV (L and %pred), TLC (L and %pred), single-breath diffusion capacity to carbon monoxide (mmol/(min kPa) and %pred)
6-minute walking test | 6 months
  Difference in change in the distance (m) walked from baseline to six months between groups in a 6-minute walking test
Blood samples | 6 months
  Difference in change from baseline to six months between groups in exercise-induced cytokine responses (interleukin-6 (pg/mL), tumour necrosis factor-α (pg/mL), C-reactive protein (μg/mL), interleukin-8 (pg/mL), and interleukin-10 (pg/mL))
Mean bolus transit time (s) (supine rest) | 6 months
  Difference in change from baseline to six months between groups in mean bolus transit time (s) (supine rest)
Mean bolus transit time (s) (adenosine infusion) | 6 months
  Difference in change from baseline to six months between groups in mean bolus transit time (s) (adenosine infusion)
Global coronary flow reserve (mL/min) | 6 months
  Difference in change from baseline to six months between groups in global coronary flow reserve (mL/min)
Pulmonary blood volume reserve (mL) | 6 months
  Difference in change from baseline to six months between groups in pulmonary blood volume reserve (mL)
Left ventricular ejection fraction (%) | 6 months
  Difference in change from baseline to six months between groups in left ventricular ejection fraction (%)
Cardiac output (L/min) (supine rest) | 6 months
  Difference in change from baseline to six months between groups in cardiac output (L/min) (supine rest)
Cardiac output (L/min) (adenosine infusion) | 6 months
  Difference in change from baseline to six months between groups in cardiac output (L/min) (adenosine infusion)
Total plasma volume | 6 months
  Difference in change from baseline to six months between groups in total plasma volume
Red blood cells | 6 months
  Difference in change from baseline to six months between groups in red blood cells
Coronary calcium score | 6 months
  Difference in change from baseline to six months between groups in coronary calcium score
Intima-media thickness (IMT) in the common carotid artery (mm) | 6 months
  Difference in change from baseline to six months between groups in intima-media thickness (IMT) in the common carotid artery (mm)
Blood samples | 6 months
  Difference in change from baseline to six months between groups in blood samples: lipids (cholesterol (mmol/l), LDL (mmol/l), HDL (mmol/l)), HbA1C (mmol/l), HsCRP (mg/L), pro-BNP (pmol/L), and TSH (10-3 IU/L)
Resistance (Rrs, R5-R20) | 6 months
  Difference in change from baseline to six months between groups in resistance (Rrs, R5-R20) measured by IOS
Reactance (Xrs, X5) | 6 months
  Difference in change from baseline to six months between groups in reactance (Xrs, X5) measured by IOS

CONTACTS AND LOCATIONS:
Locations (1):
- Center For Physical Activity Research, Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided